CLINICAL TRIAL: NCT04211532
Title: Evaluation of the ACS-NSQIP Risk Calculator for Emergent Surgery in a Spanish Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mireia Pascua-Solé, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CSPT-CIR-MP-ACSCalc
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Complications
Keywords: Surgical risk; ACS NSQIP
MeSH Terms: conditions — Postoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgery — Surgical risk is calculated according to the surgery performed.

SUMMARY:
Nowadays, quality of life and individualised medicine are becoming more important in the everyday medical practice and surgery it is not an exception. In recent years, the interest in the improvement of the quality of surgical procedures and outcomes has increased. This quality can be improved by assessing the surgical or operative risk by evaluating the postoperative mortality and morbidity.

Most of the risk stratification tools are used in elective surgery. Only few have been specifically validated for immediate or urgent. However, there are different situations. In elective interventions, the patient and the surgeon can discuss the advantages and drawbacks and postpone the decision. Moreover, an improvement in the physical status of the patient can be performed whereas in immediate or urgent surgery there is no time to neither of them.

POSSUM is used as the main tool for the prediction of mortality and morbidity and for assessing the quality care of the General Surgery Unit of Corporació Sanitària Parc Taulí. Nevertheless, this system has its limitations. It overestimates mortality in low risk patients and it does not take into account the specific surgical procedure.

That is why, it is believed that the ACS-NSQIP risk calculator -created in 2013- is a potential good tool to stratify surgical risks. In contrast with POSSUM, it considers any surgical procedure -according to the Current Procedural Terminology.

The calculator has been externally validated in population of North-America which requires emergent surgery with a somewhat underestimation of the risk. As populations have different profiles and there are different levels of care, it is needed the external validation in other countries.

In essence, there is a need of validation of risk calculators in different populations and emergency surgery (immediate and urgent) is distinct from the elective operation, therefore they should be considered separately when risk is calculated.

Therefore, there is a need of validation of the ACS NSQIP risk calculator in Spanish population which requires emergency (immediate and urgent) surgery. On the other hand, it is suggested that ACS NSQIP risk calculator performs better than POSSUM . Hence, its prediction performance is compared with POSSUM.

DETAILED DESCRIPTION:
A prospective validation cohort study is proposed. The surgical risk of the patients recruited in the study was calculated by the ACS NSQIP risk calculator and by POSSUM.

In order to compare the performance of ACS NSQIP risk calculator with POSSUM, area under the receiver operating characteristic curve (AUC) was calculated for each tool. The statistical differences between the two AUC curves were compared using P value. Calibration of the agreement between observed and predicted outcomes was tested using the Brier score. The Brier score ranges from 0 to 1. The closer the score is to 0, the more accurate is the risk prediction model.

There is a need of validation of the ACS NSQIP risk calculator in Spanish population which requires emergency (immediate and urgent) surgery. Besides, it is suggested that ACS NSQIP risk calculator performs better than POSSUM. Hence, its prediction performance is compared with POSSUM.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited were aged 18 years and older.
* Those who underwent emergency (immediate and urgent) surgery in Hospital Universitari Parc Taulí from June 2019 to June 2020.

Exclusion Criteria:

* Patients who activated of the polytraumatic code.
* Patients with proctologic disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who underwent emergent surgery is going to be recruited in the study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
ACS NSQIP outcomes | 30 days
  Each probability of the different outcomes calculated and described by the ACS NSQIP. These outcomes are the probability of suffering from: serious complication, any complication, pneumonia, cardiac complication, surgical site infection, urinary tract infection, venous thromboembolism, renal failure, ileus, anastomotic leak, return to operating room, discharge to post-acute care and death.
POSSUM outcomes | 30 days
  Each probability of the different outcomes calculated by POSSUM. These outcomes are the probability of suffering from the outcomes described for ACS NSQIP.

CONTACTS AND LOCATIONS:
Locations (1):
- Mireia Pascua Solé, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Did we prioritize quality improvement in general surgery: Time for a focus on outcomes and enhanced recovery care plans. Am J Surg. 2019 Mar;217(3):539-540. doi: 10.1016/j.amjsurg.2018.12.049. No abstract available. PMID 30777277
- [Background] Copeland GP, Jones D, Walters M. POSSUM: a scoring system for surgical audit. Br J Surg. 1991 Mar;78(3):355-60. doi: 10.1002/bjs.1800780327. PMID 2021856
- [Background] Havens JM, Columbus AB, Seshadri AJ, Brown CVR, Tominaga GT, Mowery NT, Crandall M. Risk stratification tools in emergency general surgery. Trauma Surg Acute Care Open. 2018 Apr 29;3(1):e000160. doi: 10.1136/tsaco-2017-000160. eCollection 2018. PMID 29766138
- [Background] Bilimoria KY, Liu Y, Paruch JL, Zhou L, Kmiecik TE, Ko CY, Cohen ME. Development and evaluation of the universal ACS NSQIP surgical risk calculator: a decision aid and informed consent tool for patients and surgeons. J Am Coll Surg. 2013 Nov;217(5):833-42.e1-3. doi: 10.1016/j.jamcollsurg.2013.07.385. Epub 2013 Sep 18. PMID 24055383